CLINICAL TRIAL: NCT03871400
Title: Comparison of Early Fusion Using a NanoMetalene® Implant Versus Both PEEK and Allograft Implants in Anterior Cervical Discectomy and Fusion (ACDF) With OsteoStrand™ Demineralized Bone Fibers
Brief Title: The NanoStrand Clinical Study
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Study halted prematurely and will not resume; participants are no longer receiving intervention due to coronavirus pandemic and unexpected enrollment delays.
Sponsor: SeaSpine, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: SS-NM-1801
Record Dates: First submitted 2019-03-08; First posted 2019-03-12 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Disc Degeneration;Cervical
MeSH Terms: interventions — Gene Fusion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NanoMetalene/PEEK (Other)
  Interventions: Procedure: Anterior cervical discectomy and fusion
- NanoMetalene/Allograft (Other)
  Interventions: Procedure: Anterior cervical discectomy and fusion

INTERVENTIONS:
Procedure: Anterior cervical discectomy and fusion — primary, 2-level, contiguous

SUMMARY:
A prospective, multi-center, randomized, self-controlled, single-blinded, clinical study evaluating the NanoMetalene implant as compared to the PEEK and allograft implants in ACDF for the treatment of cervical degenerative disc disease (DDD).

DETAILED DESCRIPTION:
PEEK: Polyetheretherketone ACDF: Anterior cervical discectomy and fusion

ELIGIBILITY:
Inclusion Criteria:

* Cervical degenerative disc disease
* Requires primary spinal fusion from C3-C7
* Minimum of 6 weeks of non-operative treatment
* Signed informed consent form

Exclusion Criteria:

* Uncontrolled type I or II diabetes mellitus
* Morbid obesity
* Documented history of alcohol or drug abuse
* Fever or leukocytosis
* Current systemic infection
* Active malignancy and/or current chemotherapy
* Known history of osteoporosis
* Prior fusion or total disc replacement at the operative level or an adjacent level
* Infection of the operative site
* Use of implants from other systems
* Pregnancy
* Participation in another research study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-11-18 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2021-01-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of cervical spinal levels for NanoMetalene vs PEEK interbody implants that have achieved fusion as determined by Computed Tomography (CT) analysis | 12 months
  Proportion of cervical spinal levels for NanoMetalene vs PEEK interbody implants that have achieved fusion as determined by Computed Tomography (CT) analysis

SECONDARY OUTCOMES:
Secondary CT Analysis: PEEK | 12 months
  Proportion of cervical spinal levels for NanoMetalene vs PEEK interbody implants that have achieved fusion as determined by Computed Tomography (CT) analysis
Secondary CT Analysis: Allograft | 12 months
  Proportion of cervical spinal levels for NanoMetalene vs Allograft implants that have achieved fusion as determined by Computed Tomography (CT) analysis
Secondary X-Ray Analysis | 24 months
  Proportion of cervical spinal levels for NanoMetalene vs PEEK and Allograft implants that have achieved fusion as determined by x-ray analysis
Clinical Outcomes: NDI | 24 months
  Improvement of clinical outcomes (NDI) for all enrolled patients. Improvement is a reduction of scores for all clinical outcomes. Results will be shown as change from baseline to 24 month follow-up.
  The NDI is an index derived from the Neck Disability Index Pain Questionnaire used by surgeons, clinicians and researchers to quantify disability for neck pain. Scores are from 0-100 and a lower score represents a better score.
Clinical Outcomes: VAS Arm | 24 months
  Improvement of clinical outcomes (VAS Arm) for all enrolled patients. Improvement is a reduction of scores for all clinical outcomes. Results will be shown as change from baseline to 24 month follow-up.
  The visual analogue scale (VAS) is a commonly used outcome measure for research studies. It is presented as a 100-mm horizontal line on which the patient's pain intensity is represented by a point between the extremes of "0"/no pain at all" and "100/worst pain imaginable." The study in this scale is used for the worst arm pain. A lower score represents a better score.
Clinical Outcomes: VAS Neck | 24 months
  Improvement of clinical outcomes (VAS Neck) for all enrolled patients. Improvement is a reduction of scores for all clinical outcomes. Results will be shown as change from baseline to 24 month follow-up.
  The visual analogue scale (VAS) is a commonly used outcome measure for research studies. It is presented as a 100-mm horizontal line on which the patient's pain intensity is represented by a point between the extremes of "0"/no pain at all" and "100/worst pain imaginable." The study in this scale is used for neck pain. A lower score represents a better score.

CONTACTS AND LOCATIONS:
Overall Officials: Khalid Abbed, MD, Principal Investigator — Yale University
Locations (11):
- United States (11):
  - Barrow Brain and Spine, Phoenix, Arizona
  - University of California, San Diego, La Jolla, California
  - University of Southern California, Los Angeles, California
  - UCLA Health, Santa Monica, California
  - University of Colorado Hospital, Aurora, Colorado
  - Spine Colorado, Durango, Colorado
  - Emory, Atlanta, Georgia
  - Hughston Clinic, Columbus, Georgia
  - Northwestern University, Chicago, Illinois
  - OrthIndy, Indianapolis, Indiana
  - Henry Ford, Jackson, Michigan

IPD SHARING:
Plan to Share IPD: No